CLINICAL TRIAL: NCT05982210
Title: The Influence of the Diaphragm Muscle and Pain Perception on Lower Limb Neuromuscular Control Parameters in Sports Practice: Application of Breathing Exercises and Manual Therapy of the Diaphragm Muscle and Ribs Protocol
Brief Title: The Influence of the Diaphragm Muscle and Pain Perception on Lower Limb Neuromuscular Control in Sports Practice.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Imma Vergara Busquets, PhD Student, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FIS-2022-13
Record Dates: First submitted 2023-07-29; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Diaphragm; Relaxation
Keywords: Core Stability; Diaphragm Muscle; Rib Cage; Breathing Biomechanics
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The Control Group does not have any interventions applied.
- Intervention Group (Experimental): The Intervention Group will take part in the experimental process. A clinical practice protocol about breathing exercises and diaphragm and ribs manual therapy will be applied, in a total duration of 15 minutes, twice a week during eight weeks.
  Interventions: Other: Breathing Exercises and Manual Therapy of the Muscle Diaphragm and Ribs Protocol

INTERVENTIONS:
Other: Breathing Exercises and Manual Therapy of the Muscle Diaphragm and Ribs Protocol — The intervention consists on applying a protocol based on five different exercises, compound by breathing exercises and manual therapy of the muscle diaphragm and the ribs, applied by a physiotherapist.
  Arms: Intervention Group

SUMMARY:
Core stability is maintained mainly by muscle function of abdominal and lumbar region, including the diaphragm muscle. It is known that exists a connection between trunk's muscle activity and the movement of lower limb and lower limb and low back injuries are related to core alterations. Thus, a randomized clinical trial is planned to analyze the effectiveness of an exercises and manual therapy of the diaphragm and ribs program designed, aiming to analyze the correlation between rib cage mobility and lower limb neuromuscular control in young healthy subjects.

DETAILED DESCRIPTION:
The aim of the study consists on analysing the correlation between rib cabe mobility and neuromuscular control parameters of lower limb, as well as pain perception in young healthy adults sports players. A clinical practice protocol consisting on breathing exercises and manual therapy of the muscle diaphragm and the ribs will be applied twice a week during eight weeks. As a result, could be an increasement of the neuromuscular control parameters, described with the outcome measures of rib cage mobility, lower limb power and stability, and pain perception. If the results stablish correlation between the rib cage mobility and neuromuscular control parameters of lower limb, could be helpful in healthcare and sports science field in order to take in account the diaphragm biomechanics when treating lower limb injuries and facing its prevention.

ELIGIBILITY:
Inclusion Criteria:

* Physical Activity Practice: at least 150-300min of moderate activity or 75-100min of intense aerobic activity, twice a week.
* Physical activity or sports practice involve mostly lower limb muscles activation.
* Core Stability exercises least twice a week. Includes at least 3 of the 6 exercises listed: bridge exercises, standard plank, lateral plank, superman exercise, mountain climber and plank variations.

Exclusion Criteria:

* Musculoskeletal injury currently or in the past 6 months.
* Abdominal or thoracic surgery.
* Nervous System disease.
* Hiatal Hernia or visceral disease.
* Pelvic floor alterations or disease.
* Breathing restrictions: disease or infection, asthma, anxiety or other non controlled alterations.
* Treatment of the diaphragm muscle the past 6 months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Rib Cage Mobility | Week 0, Week 4 and Week 9
  The the rib cage mobility is assessed using a measuring tape. The measuring tape assess the diameter of the rib cage between a maximal inspiration and maximal expiration. Two anatomical marks are described: the superior mark is formed by the third intercostal space, de clavicular line and spinous apophysis of the thoracic vertebra number five; and the inferior mark is formed by xiphoid process and the spinous apophysis of the thoracic vertebra number ten.
  The subjects stand with the hands on the head and the evaluator mantains the measuring tape around the rib cage of the subject. The subject inhales by the nose expanding the lungs and exhales by the mouth until the lungs are empty. The measures are taken three times, at the beginning of each inspiratory and expiratory cycle.
  The repetition is failed if the subject makes an apnea or cough.

SECONDARY OUTCOMES:
Lower Limb Power | Week 0, Week 4 and Week 9
  My Jump Lab App is used to asses lower limb power through jump analysis. The device is fixed with a tripod, 50 centimetres away from the floor, focused on the frontal plane of the subject. The subject makes a CounterMovement Jump (CMJ) which is recorded in 240 frames/second. The subject is standing with shoes and knees extended and the hands on the hips. From this position, the subject quickly makes a knee flexion until 90 degrees followed by a quick knee extension before taking a maximum vertical jump.
  After de jump is recorded, the take off frame and the landing frame are indicated in the app, and calculates automatically the power of lower limb.
  Three repetitions are recorded from each lower limb.
Lower Limb Stability | Week 0, Week 4 and Week 9
  The Star Excursion Balance Test (SEBT) is used to assess lower limb stability. Three tape strips are placed on the floor: anterior (A), posteromedial (PM) and posterolateral (PL), leaving 120 degrees angulation between A and PM/PL, and 90 degrees between PM and PL, converging at the 0 mark.
  The participant stands in monopodal position with hands on the hips, without shoes or socks. The anterior part of the foot stays in the 0 mark for the A direction, and the heel por PM and PL. The participant slides the free foot through the tape without touching it until reaching the maximum distance, registrated in centimeters. The repetition is failed if the participant touches the floor, move the baseline foot or touches the tape more than once.
  Three repetitions will be recorded for each lower limb and for each direction. The length of the lower limb is measured with the distance between the anterosuperior iliaca spine and the external tibial malleolus.
Pain Perception | Week 0, Week 4 and Week 9
  The Numeric Rating Scale (NRS) is used to assess pain perception. The NRS is a visual scale composed by 11 different numeric points, within the 0 represents inexistent pain and the 10 represents the maximal pain imaginable.
  The subject indicates which number adjusts to the pain intensity experimented related to the lower limb.

CONTACTS AND LOCATIONS:
Overall Officials: María Caridad Bagur, Study Director — Universitat Internacional de Catalunya; Xantal Borràs, Study Director — Universitat de Vic
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No